CLINICAL TRIAL: NCT07131046
Title: A Comparative Analysis of Combined Superficial Cervical Plexus and Supraorbital Blocks Compared to Scalp Blocks During Craniotomy: a Review of Opioid Consumption and The Suppression of Hemodynamic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, Anesthesiologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes1002
Record Dates: First submitted 2025-07-28; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Craniotomy Surgery; Regional Anaesthesia; Scalp Block; Plexus Block;Analgesia;Neurosurgery
Keywords: superficial cervical plexus block; supraorbital nerve block; scalp block; craniotomy; remifentanil; regional anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of superficial cervical plexus block and supraorbital block (Experimental)
  Interventions: Procedure: Combination of superficial cervical plexus block and supraorbital block
- Scalp block (Sham Comparator)
  Interventions: Procedure: Scalp block with bupivacaine alone

INTERVENTIONS:
Procedure: Combination of superficial cervical plexus block and supraorbital block — The combined anaesthesia technique involves the use of general anaesthesia and regional block in the superficial cervical plexus and supraorbital areas, with 6 ml of 0.25% bupivacaine injected into the superficial cervical plexus area and 2 ml into the supraorbital area.
  Arms: Combination of superficial cervical plexus block and supraorbital block
Procedure: Scalp block with bupivacaine alone — A combination anaesthesia technique is used that involves general anaesthesia and scalp block. Scalp block using 0.25% bupivacaine in the supraorbital area (2 ml), supratrochlear (2 ml), zygomaticotemporal (2 ml), auriculotemporal (2 ml), major occipital (2 ml) and minor occipital (2 ml).
  Arms: Scalp block

SUMMARY:
Perioperative pain management in craniotomy requires the administration of effective regional anesthetic techniques to reduce the use of systemic opioids and optimize hemodynamic control. Scalp block has been demonstrated to suppress hemodynamic response; however, its implementation generally involves a large number of injection points (six nerves that must be blocked bilaterally, resulting in a total of 12 injection points) and the possibility that not all nerve points are adequately blocked. Meanwhile, superficial cervical plexus and supraorbital block involves fewer injection points (two nerves to be blocked bilaterally, for a total of four injection points) with an analgesia area that may be sufficient to facilitate craniotomy surgery, including the insertion of Mayfield pins, consisting of only three pins, where the pin insertion area is not too large. The objective of this study is to compare the efficacy of combined superficial cervical plexus and supraorbital block with scalp block in reducing intraoperative opioid consumption and controlling hemodynamic response in craniotomy surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been scheduled to undergo a craniotomy procedure that has been deemed medically necessary and electively scheduled. The aforementioned procedure will be performed under the administration of general anesthesia and the utilization of Mayfield pins.
2. Adult patients who have reached an age of 18 years and have not yet reached 65 years of age are included in this study.
3. Patients with ASA classification 1 - 3
4. The patient has expressed their willingness to participate in a research study and has provided their signature on an informed consent form.

Exclusion Criteria:

1. The patient has been diagnosed with an infection in the area where the block needle insertion is to be performed.
2. The subjects of this study were patients with a body mass index (BMI) greater than 30 kg/m2 who were classified as Grade II obese.
3. The patient is currently undergoing treatment with a beta-blocker.
4. Patients in whom intraoperative evoked potential monitoring is scheduled.
5. The patient is scheduled to undergo a total intravenous anesthesia technique
6. The history of an allergy to local anesthesia is presented before.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Remifentanil consumption for each step of surgery | intraoperative
  The target effect of the highest dose of Remifentanil administered by total controlled infusion when there is an increase in MAP or heart rate by more than 20% of the initial value for 30 seconds during Mayfield pin placement, skin incision, periosteal manipulation, and skin suturing.
The total amount of Remifentanil administered during the operation | Intraoperative
  The total amount of remifentanil that the medical team used during the surgery
The greatest alterations in mean arterial pressure (MAP) during the pinning procedure, followed by skin incision, periosteum manipulation, and skin suture. | Intraoperative
  Changes in mean arterial pressure were measured at several points: 30 minutes after the block was administered; during pin insertion; during skin incision; during periosteal incision; and during skin suturing.
The greatest alteration in heart rate during the pinning procedure, followed by skin incision, periosteum manipulation, and skin suture. | Intraoperative
  Changes in heart rate were measured at several points: 30 minutes after the block was administered; during pin insertion; during skin incision; during periosteal incision; and during skin suturing.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangungkusoma Central Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sato T, Nishiwaki K. Accuracy of landmark scalp blocks performed during asleep-awake-asleep awake craniotomy: a retrospective study. JA Clin Rep. 2021 Jan 9;7(1):8. doi: 10.1186/s40981-021-00412-4. No abstract available. PMID 33420848
- [Background] Girard F, Quentin C, Charbonneau S, Ayoub C, Boudreault D, Chouinard P, Ruel M, Moumdjian R. Superficial cervical plexus block for transitional analgesia in infratentorial and occipital craniotomy: a randomized trial. Can J Anaesth. 2010 Dec;57(12):1065-70. doi: 10.1007/s12630-010-9392-3. Epub 2010 Sep 28. PMID 20878375
- [Background] 1. Department of Neurology, Faculty of Medicine, Universitas Indonesia/Rumah Sakit Cipto Mangunkusumo, Jakarta, Indonesia, Aninditha T. Adults brain tumor in Cipto Mangunkusumo General Hospital: A descriptive epidemiology. Ro J Neurol. 31 Desember 2021;20(4):480-4.